CLINICAL TRIAL: NCT04594057
Title: The Impact of Vestibular Rehabilitation on the Longitudinal Recovery of Laboratory, Clinical, and Community-Based Measures of Head and Trunk Control in People With Acquired Vestibulopathy
Brief Title: Longitudinal Recovery of Laboratory, Clinical, and Community-Based Measures of Head and Trunk Control in People With Acquired Vestibulopathy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty with enrollment secondary to COVID
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IRB_00125069; NIFTI (Other Grant/Funding Number: Foundation for Physical Therapy)
Record Dates: First submitted 2020-09-11; First posted 2020-10-20 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2020-10

CONDITIONS: Vestibular Schwannoma; Vestibular Disorder
MeSH Terms: conditions — Neuroma, Acoustic; Vestibular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Start (Active Comparator): Begin 6 weeks of gaze and postural stability training 10-14 days following surgery.
  Interventions: Behavioral: Gaze and Postural Retraining Exercise
- Delayed Start (Experimental): Begin 6 weeks of gaze and postural stability training 6 weeks following surgery.
  Interventions: Behavioral: Gaze and Postural Retraining Exercise

INTERVENTIONS:
Behavioral: Gaze and Postural Retraining Exercise — Gaze and Postural Stability The duration and content of the Gaze and Postural Stability (GPS) intervention is specifically designed to focus on gradually increasing difficulty of gaze and postural stability exercises.
  The target duration of each in clinic visit will be 90 min (15 min of gaze stability exercises, 15 min of postural stability exercises and approximately 60 min for the standard care control intervention with rest interspersed throughout the exercise session.
  Gaze stability exercise will consist of progressive Vestibular-occular training.
  Postural stability exercises will consist of progressive static and dynamic postural training.

SUMMARY:
This study is designed to examine the true impact inner-ear dysfunction has on patient head movement kinematics, activity levels, and participation, and (2) to explore the efficacy of rehabilitation on laboratory, clinical, and community-based outcomes in people following surgical removal of a schwannoma from the inner-ear nerve.

DETAILED DESCRIPTION:
In this project we will focus on characterizing deficits in community-based performance (i.e., head and trunk control during simulated community activities, short term community mobility, and patient reported participation) and relating these deficits to laboratory (i.e., video head impulse testing and corrective postural responses) and clinical (i.e., MiniBEST and dynamic visual acuity, and visual spatial cognition) measures of gaze and postural stability in individuals with varied forms of vestibulopathy (unilateral vestibular neuritis, bilateral vestibular loss, migraine related vestibulopathy, concussion, BPPV, Multiple Sclerosis). Additionally, we will examine the longitudinal change of laboratory, and community-based measures of gaze and postural in two cohorts of people with a specific form of unilateral vestibular loss (Vestibular Schwannoma resection); one group of these individuals will receive 6 weeks of vestibular rehabilitation during the acute onset of symptoms and the other one will begin intervention 6 weeks post onset. This portion of the proposed project will test my global hypothesis that changes in community-based performance of head and trunk control impair recovery following the onset of VH.

Aim 1: In individuals with vestibulopathy, characterize and compare laboratory and clinical measures of body structure, function, and performance to community-based, activity levels, performance, and patient reported participation. Hypothesis 1: The severity of laboratory and clinically measured gaze and postural stability function deficits will not strongly correlate with head and trunk control during community-based performance or patient reported participation. Hypothesis 2: The nature and severity of laboratory and clinically measured gaze and postural stability function deficits will differ between varied diagnostic groups.

Aim 2: In individuals with unilateral vestibular hypofunction following unilateral vestibular schwannoma resection, examine the longitudinal trajectories of laboratory and clinical measures of body structure, function and performance, and community-based performance, activity levels, and patient reported participation during periods of spontaneous and rehabilitation driven recovery. Hypothesis: Recovery of laboratory and clinical measures will follow different trajectories than measures of community-based performance and patient reported participation during both periods of spontaneous and rehabilitation driven recovery.

ELIGIBILITY:
Inclusion Criteria:

* Reports of dizziness as indicated by Dizziness handicap inventory score >0
* Undergoing a vestibular schwannoma resection surgery and/or vestibular hypofunction diagnosed using bedside examination
* Able to perform community ambulation

Exclusion Criteria:

* Presence of cardiovascular, orthopedic, or other neurologic diagnosis that limits ability to complete study testing, or causes other forms of dizziness.
* Blindness
* Peripheral neuropathy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-12-10 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Dizziness Handicap Inventory (DHI) | Change baseline to 6 weeks
  Dizziness Handicap Inventory (DHI): The DHI is a self assessment inventory designed to evaluate the self-perceived handicap effects imposed by dizziness or unsteadiness and has documented test-retest and internal consistency reliability in PwMS. The DHI consists of 25 questions subgroup into functional, emotional, and physical components. The total score ranges from 0-100, with higher scores indicating greater handicap. Change from baseline to 6 weeks post surgery.
Change in miniBEST test | Change from baseline to 6 weeks
  the 14-item Mini-BESTest which includes four sections (anticipatory postural adjustments, reactive postural responses, sensory orientation, and stability in gait) relevant to postural control and stability in MS. The maximum possible score is 28 with higher scores indicating better balance. Tasks within the Mini-BEST test require head and/ or body motion, which will be assessed using body-worn 3D accelerometers. The Change from the baseline score to the 6 weeks post surgery score.
Change in Community-simulated Ambulatory Task (CAT) | Change from Baseline to 6 weeks
  Community-simulated walking task consisting of turns, stairs, and inside/outside ambulation requiring specific use of head and trunk turns. Change from baseline to 6 weeks post surgery.
Change in Passive Angular Vestibular Reflex Testing | Change from Baseline to 6 weeks
  The angular vestibular ocular reflex (aVOR) gain will be calculated as the ratio of the de-saccaded eye velocity Area Under the Curve (AUC) over the head velocity AUC between the onset of the head impulse to the moment when head velocity returns to zero. Change from baseline to 6 weeks post surgery in aVOR gain.

SECONDARY OUTCOMES:
Activities Balance Confidence Scale (ABC) | Baseline, 10 days post surgery, 6 weeks, and 12 weeks post surgery.
  The Activity Specific Balance Confidence Scale (ABC) is a 16-item self-reported measure of balance confidence in performing various activities of daily living. Each question requires an individual to grade his or her self on a scale of 0 to 100 percent for their level of confidence and higher scores indicate greater balance confidence in performing these activities.
Life Space Assessment | Baseline, 10 days post surgery, 6 weeks, and 12 weeks post surgery.
  The Life Space Assessment is self-report questionnaire that captures the amount of time which a person interacts with differing levels of their environment.
Dynamic Visual Acuity | Baseline, 10 days post surgery, 6 weeks, and 12 weeks post surgery.
  The Dynamic Visual Acuity (DVA) test is a valid and reliable functional measure of gaze stability that utilizes head rotations representing natural head velocities during daily activities. The variable logMAR is the standard measurement for DVA and is equal to log10x, where x is the minimum angle resolved, in arcmin, with 1 arcmin equal to 1/60°). The better one's visual acuity, the lower one's logMAR score.
Compensatory Saccade Frequency | Baseline, 10 days post surgery, 6 weeks, and 12 weeks post surgery.
  The number of Compensatory Saccades (CS) per Head Rotation (CS/HR) will be manually counted per head rotation. Collected at intervention completion and 1-month follow-up adjusting for baseline (values collected at baseline assessment).
Daily Step Activity | Baseline, 10 days post surgery, 6 weeks, and 12 weeks post surgery.
  Step activity monitors will be used to quantify daily step activity during over a 4 day window.
Postural Sway | Baseline, 10 days post surgery, 6 weeks, and 12 weeks post surgery.
  The amount of postural sway during quiet stance on firm, foam, and incline surfaces will be assessed using 3D accelerometers.
Modified Physical Performance Test (mPPT) | Baseline, 10 days post surgery, 6 weeks, and 12 weeks post surgery.
  The mPPT assess basic and complex activities of daily living including rising from a chair, picking an object up from the floor, donning and doffing a jacket, placing an item on a shelf, a 50 foot walk, 360 degree turns, and ascending an descending stairs.
Repeated Battery of the Assessment of Neuropsychological Status (RBANS): Line Orientation Sub-Test | Baseline, 10 days post surgery, and 12 weeks post surgery.
  A test of visual spatial cognition that requires the participant to try and correctly identify the orientation of two lines presented to them with 12 other line options. Scores range from 0-20 based on correctness of line orientation on 10 different trials.
Repeated Battery of the Assessment of Neuropsychological Status (RBANS): Figure Copy Sub-Test | Baseline, 10 days post surgery, and 12 weeks post surgery.
  A test of visual spatial cognition that requires the participant to copy a multiple shape figure and is scored from 0-20 based on the correctness of the figure copy.

OTHER OUTCOMES:
Two-Minute Walk (2MWT) | Baseline, 10 days post surgery, 6 weeks, and 12 weeks post surgery.
  The distance walked in 2 minutes (Two-Minute Walk [2MWT]) is a valid and reliable measure of locomotor ability in populations with a variety of chronic diseases. Higher values reflect greater ability.
Visual Analog Scale of Dizziness | Baseline, 10 days post surgery, 3 weeks, 6 weeks, 9 weeks, and 12 weeks post surgery.
  A single mark will be made along a 10 cm line indicating the amount of dizziness experienced ranging from "no dizziness" to "worst possible dizziness".
Visual Analog Scale of Unsteadiness | Baseline, 10 days post surgery, 3 weeks, 6 weeks, 9 weeks, and 12 weeks post surgery.
  A single mark will be made along a 10 cm line indicating the amount of unsteadiness experienced ranging from "no unsteadiness" to "worst possible unsteadiness".

CONTACTS AND LOCATIONS:
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No